CLINICAL TRIAL: NCT04844840
Title: A Phase 2, Multi-Center, Randomized, Multiple Arm, Controlled Pilot Study to Evaluate the Safety and Efficacy of Various Doses of STP705 in Reducing Post- Keloidectomy Keloid Recurrence
Brief Title: A Study for Safety and Efficacy Evaluation of Various Doses of STP705 in Reducing Keloid Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SRN-705-007
Record Dates: First submitted 2021-04-08; First posted 2021-04-14 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — Injections

STUDY DESIGN:
Intervention Model Description: 10 subjects each will be randomly allocated to either the assigned STP705 treatment group, placebo or SOC alone in a 1:1:1:1:1:1 ratio.
  An individual, independent of the clinical trial team, will develop the randomization schedules. The actual randomization assignment will be prepared through a web-based system. STP705 or placebo will be injected intradermally at the keloid excision site.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. All subjects, investigator, and site staff (except unblinded pharmacist or designated site staff) in the study will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: STP705 10 μg dose (Experimental): STP705 at the assigned dose will be injected intradermal into the excised keloid site
  Interventions: Drug: STP705
- Cohort 2: STP705 20 μg dose (Experimental): STP705 at the assigned dose will be injected intradermal into the excised keloid site
  Interventions: Drug: STP705
- Cohort 3: STP705 30 μg dose (Experimental): STP705 at the assigned dose will be injected intradermal into the excised keloid site
  Interventions: Drug: STP705
- Cohort 4: STP705 40 μg dose (Experimental): STP705 at the assigned dose will be injected intradermal into the excised keloid site
  Interventions: Drug: STP705
- Cohort 5: Placebo control (Placebo Comparator): Placebo (saline) will be injected intradermal into the excised keloid site
  Interventions: Other: Placebo
- Cohort 6: SOC alone (No Intervention): SOC (no injection)

INTERVENTIONS:
Drug: STP705 — STP705 is composed of two siRNA oligonucleotides, targeting TGF-β1 and COX-2 mRNA, respectively
  Other Names: STP705 Powder for Injection
  Arms: Cohort 1: STP705 10 μg dose; Cohort 2: STP705 20 μg dose; Cohort 3: STP705 30 μg dose; Cohort 4: STP705 40 μg dose
Other: Placebo — Saline
  Arms: Cohort 5: Placebo control

SUMMARY:
Phase 2, randomized, double-blind, multiple arm, controlled study to evaluate safety & efficacy of various doses of STP705 in reducing post Keloidectomy keloid recurrence.

DETAILED DESCRIPTION:
The objective of this study isto assess the safety, tolerability, and efficacy of various doses of STP705 and placebo via intradermal injection into the keloid excision site, to prevent the recurrence of keloids following their excision.

A total of up to 60 adult subjects will be enrolled. One eligible qualifying keloid will be excised. The subjects will be randomized to receive STP705, placebo or SOC alone (no injection) for treatment of the keloidectomy excision suture line.

To be eligible, keloid scar(s) must have been present for at least one year with a target keloid area on the trunk or extremity (non-peri-orbital/-anogenital/-scalp), measures ≥0.30cm2, and be suitable for surgical excision which will result in a single wound no greater than 7cm long.

The study is divided into 3 phase: screening phase (4 weeks), Treatment phase (up to 4 weeks +/- allowed windows), Follow up phase (up to 52 weeks +/- allowed windows).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age, inclusive having at least one keloid scar.
2. Female subjects of child-bearing potential must agree to the use of an effective method(s) of contraception beginning at or before the screening visit until one month after administration of the final study dose. For the purposes of the protocol, highly effective method(s) of contraception will be defined as consistently and correctly used implants, injectables, combined oral contraceptives, sexual abstinence or a vasectomized partner.
3. The keloid scar(s) must have been present for at least one year with a target keloid area on the trunk or extremity (non-peri-orbital/-anogenital/-facial/-scalp), measures ≥0.30cm2, and be suitable for surgical excision which will result in a single wound no greater than 7cm long.
4. Able and willing to give written informed consent.
5. Willing to comply with the follow up schedule for 12 months.
6. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, or vital sign abnormalities as deemed by the PI.

Exclusion Criteria:

1. Prior treatment of the keloid scar in the previous 6 weeks.
2. The keloid scar must not have undergone prior surgical excisions (laser, cryotherapy or surgery).
3. The keloid scar must not have undergone prior radiation treatment.
4. Pregnant, lactating, or planning to become pregnant during the course of the study.
5. Advanced or poorly controlled diabetes.
6. Active local infection at the treatment site and/or systemic infection that would in the opinion of the Investigator affect the treatment site.
7. Any medical or surgical condition that will interfere with required study activities or assessments or that make the study treatments contraindicated in the opinion of the study Investigator.
8. Unwilling to refrain from use of any other scar treatment therapy/scar improving product, during the study.
9. Regular, continuous use of systemic corticosteroid therapy or topical corticosteroid use in the area to be treated.
10. Current participation or participation within the last 1 months in the study of an investigational drug, device, or biologic.
11. Unable or unwilling to follow post-operative instructions.
12. Mentally or legally incapacitated or has significant emotional problems at the time of screening visit or expected during the conduct of the study.
13. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds, or drug product excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Rate of Recurrence | 12 months
  Rate of recurrence in subjects undergone surgery alone (with or without placebo) vs surgery and STP705

SECONDARY OUTCOMES:
Change of Keloid volume/size | 12 months
  Change in size of post excision keloid from baseline by volumetric measurements using quantitative imaging
Change of Keloid size | 12 months
  Change of Keloid scar appearance from baseline evaluated by caliper
Change of Keloid scar appearance | 12 months
  Change of Keloid scar appearance from baseline evaluated by POSAS
Change in DLQI score | 12 months
  The Dermatology Life Quality Index (DLQI) is a self-reported 10-item questionnaire assessing the impact of skin disease on the patient over the previous week. The items cover symptoms, treatment, activity limitations, and emotional reactions to having a skin disease. Nine items have four response options: "Not at all", "A little", "A lot", and "Very much", whereas item 7 first asks whether work or study has been prevented and then (if "No") to what degree the skin condition has been a problem at work/study ("A lot", "A little", or "Not at all"). Eight of the items also have a "Not relevant" option that is scored "0", indicating no problem. Individual item scores are summed to derive a total DLQI score that can range from 0 to 30, with higher scores indicating worse health- related quality of life (HRQL).
Change in mVSS score | 12 months
  The modified Vancouver Scar Scale (mVSS) performs a comprehensive measurement rating characteristic of pigmentation, vascularity, pliability, and height. For each subject, a total Vancouver score was determined by summing the scores of the four individual parameters to generate a score ranging from 0 to 15 points, with higher scores indicating worse score severity.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nestor, MD, Principal Investigator — Center for Clinical and Cosmetic Research; David Goldberg, MD, Principal Investigator — Schweiger Dermatology Group; Brenda LaTowsky, MD, Principal Investigator — Investigate MD
Locations (3):
- United States (3):
  - Investigate MD, Scottsdale, Arizona
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Schweiger Dermatology, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No